CLINICAL TRIAL: NCT00209573
Title: A Phase III, Randomized, Open-Label Study to Assess the Safety and Efficacy of AQUAVAN Injection Versus Midazolam HCl for Sedation in Patients Undergoing Colonoscopy Procedures
Brief Title: A Study of AQUAVAN® Injection Versus Midazolam HCl for Sedation in Patients Undergoing Elective Colonoscopy
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Eisai Inc. (Industry)
Collaborators: PPD Development, LP (Industry); Bio Analytical Research Corporation (Industry); MDS Pharma Services (Industry); Coghlan Group (Plasma Sample Supplies) (Unknown)
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 3000-0410
Record Dates: First submitted 2005-09-13; First posted 2005-09-21 (Estimated); Last update posted 2008-11-07 (Estimated); Status verified 2008-11

CONDITIONS: Colonoscopy; Colon Polyps
Keywords: Colonoscopy; Sedation
MeSH Terms: conditions — Colonic Polyps | interventions — fospropofol

INTERVENTIONS:
Drug: fospropofol disodium

SUMMARY:
This study was designed to demonstrate that AQUAVAN® is effective in providing adequate sedation in patients undergoing colonoscopy as well as to assess the safety profile of AQUAVAN versus that of midazolam. Prior to the procedure, patients received fentanyl citrate for pain management followed five minutes later by AQUAVAN® Injection for sedation. Throughout the procedure, study personnel assessed the patient's vital signs and depth of sedation. After the procedure, the patient, physician, and an evaluator were asked to complete satisfaction surveys.

DETAILED DESCRIPTION:
This is a randomized, open-label study designed to assess the safety and efficacy of AQUAVAN® Injection versus midazolam HCl following pretreatment with an analgesic, fentanyl citrate injection, in producing sedation in patients undergoing colonoscopy. Randomization will be stratified by site. Following completion of pre-procedure sedation assessments, patients will be randomly assigned to 1 of the 2 i.v. treatment groups at a 3:1 (AQUAVAN® Injection: midazolam HCl) allocation ratio. All study patients, irrespective of treatment group assignment, will receive fentanyl citrate injection as an analgesic pretreatment. Supplemental doses of fentanyl citrate injection may be administered if the patient reports pain or if inadequate analgesia is present as demonstrated by increased heart rate and/or blood pressure in the presence of adequate sedation. At no time should fentanyl citrate injection be administered to increase sedation levels. AQUAVAN® Injection and midazolam HCl will be administered to induce a state of adequate sedation, defined as a Modified Observer's Assessment of Alertness / Sedation (OAA/S) score of 4 or less. Supplemental doses will be administered to increase depth or duration of sedation. Supplemental doses will not be administered if the Modified OAA/S score is 2 or less or if there is no purposeful response to stimulation. The depth of sedation will be measured by the Modified OAA/S scale, a validated measure. Patient and Investigator assessments will be used to confirm the depth of sedation provided met the goals of sedation, reduction of anxiet, and reduced awareness.

ELIGIBILITY:
Inclusion Criteria:

* Patient provided a signed/dated Informed Consent and HIPAA authorization after receiving a full explanation of the extent and nature of the study;
* Patient, if female, were surgically sterile, postmenopausal or non-pregnant and non lactating using an acceptable method of birth control for at least 1 month prior to dosing, with a negative urine pregnancy test result at screening and predose periods; and
* Patient met American Society of Anesthesiologists (ASA) Physical Status Classification System of I to III.

Exclusion Criteria:

* Patient had a history of allergic reaction or hypersensitivity to any anesthetic agent, narcotic, or benzodiazepine;
* Patient did not meet nils per os (NPO) status per ASA Guideline or institution's guideline.
* Patient had condition(s) that, in the opinion of the Investigator, could interfere with appropriate airway management;
* Patient participated in an investigational drug study within 1 month prior to study start;
* Patient had a history of mental or visual impairment that would not permit successful measurement of cognitive evaluations;
* Patient was unwilling to adhere to pre- and postprocedural instructions; or
* Patient for whom the use of fentanyl or midazolam was contraindicated.

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270
Dates: Start 2004-09; Study Completion 2004-12 (Actual)

PRIMARY OUTCOMES:
The primary efficacy hypothesis was that AQUAVAN could sedate (≥3 consecutive Modified OAA/S scores ≤4) patients AND that they could complete the procedure successfully without requiring alternative sedative medication AND without requiring manual or

SECONDARY OUTCOMES:
Secondary Efficacy Endpoints
Time to Fully Recovered from end of procedure
Time to Fully Alert from end of procedure
Change from baseline DSST score over time during recovery period
Duration and percent of time when a patient's Modified OAA/S score is at each level between the first dose of study medications and Fully Alert, inclusive
Duration of sedation
Number of doses of study medication administered for the procedure
Time to sedation
Time to reach splenic flexure, hepatic flexure, cecum, and end of procedure
Number of repositionings
Number of procedure interruptions due to inadequate sedation
Patient's rating of experience after Fully Recovered
Patient's rating at 24 hour post discharge telephone survey
Investigator's rating at end of procedure
Blinded evaluator's rating after patient is Fully Recovered
Safety Endpoints
Nature, frequency, severity, relationship to treatment, and outcome of all adverse events
Airway assistance
Sedation-related adverse events
Laboratory parameters and vital signs
Concomitant medications

CONTACTS AND LOCATIONS:
Overall Officials: James Jones, MD,PharmD, Study Director — Eisai Inc.